CLINICAL TRIAL: NCT00002608
Title: Cisplatin, Doxorubicin and Tamoxifen in the Treatment of Incurable Soft Tissue and Endocrine Malignancies
Brief Title: Combination Chemotherapy and Tamoxifen in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Regional Cancer Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CAN-OTT-9401; CDR0000063892 (Registry Identifier: PDQ (Physician Data Query)); NCI-V94-0566
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2005-05

CONDITIONS: Adrenocortical Carcinoma; Brain and Central Nervous System Tumors; Head and Neck Cancer; Liver Cancer; Malignant Mesothelioma; Pheochromocytoma; Sarcoma
Keywords: childhood brain tumor; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent adult soft tissue sarcoma; recurrent childhood brain tumor; childhood liver cancer; stage IV childhood liver cancer; recurrent childhood liver cancer; advanced malignant mesothelioma; recurrent malignant mesothelioma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; recurrent adult brain tumor; stage IV adrenocortical carcinoma; recurrent adrenocortical carcinoma; stage IV papillary thyroid cancer; stage IV follicular thyroid cancer; thyroid gland medullary carcinoma; anaplastic thyroid cancer; recurrent thyroid cancer; adult brain stem glioma; adult medulloblastoma; adult glioblastoma; metastatic pheochromocytoma; recurrent pheochromocytoma; childhood soft tissue sarcoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; adult anaplastic astrocytoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult pilocytic astrocytoma; adult subependymoma; recurrent childhood brain stem glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood ependymoma; stage IV adult soft tissue sarcoma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; adult diffuse astrocytoma
MeSH Terms: conditions — Adrenocortical Carcinoma; Central Nervous System Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Mesothelioma, Malignant; Pheochromocytoma; Sarcoma; Carcinoma, Hepatocellular; Brain Neoplasms; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Carcinoma, Medullary; Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms; Medulloblastoma; Glioblastoma; Astrocytoma; Oligodendroglioma; Ependymoma; Glioma; Glioma, Subependymal; Optic Nerve Glioma; Familial ependymoma; Gliosarcoma | interventions — Cisplatin; Doxorubicin; Tamoxifen; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: tamoxifen citrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. Estrogen can stimulate the growth of tumor cells. Hormone therapy using tamoxifen may fight cancer by blocking the uptake of estrogen. Combining tamoxifen with chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cisplatin and doxorubicin together with tamoxifen works in treating patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and efficacy of cisplatin, doxorubicin, and tamoxifen (CAT) in patients with soft tissue sarcoma, glioma, mesothelioma, hepatoma, thyroid cancer, or adrenal cancer.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive cisplatin IV over 1-2 hours followed immediately by doxorubicin IV over 15-30 minutes on days 1-3 and oral tamoxifen twice daily on days 4-17. Treatment continues every 3 weeks in the absence of the total cumulative doxorubicin dose reaching at least 500 mg/m2, disease progression, or unacceptable toxicity. Patients who achieve partial remission (PR) undergo local surgery or radiotherapy, if feasible, to convert PR to complete remission.

Patients are followed every 2 months for 1 year and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven soft tissue sarcoma, glioma, mesothelioma, hepatoma, thyroid cancer, or adrenal cancer with clinical, radiological, or histologic evidence of incurability
* Patients with thyroid cancer must have failed radioactive iodine
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 65 and under

Performance status:

* ECOG 0-2

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 140,000/mm3

Hepatic:

* Bilirubin normal

Renal:

* Creatinine less than 1.47 mg/dL

Cardiovascular:

* Left ventricular ejection fraction at least 50% by MUGA scan
* No congestive heart failure
* No severe, uncontrolled hypertension
* No ischemia, life-threatening arrhythmia, or conduction disturbance by ECG

Other:

* No allergy to study medications
* No uncontrolled infection
* No active abuse of ethanol that would preclude treatment
* No other prior or concurrent malignancy
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 1 prior chemotherapy regimen
* No prior anthracycline or cisplatin
* At least 3 weeks since other prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to more than 25% of bone marrow
* At least 3 weeks since other prior radiotherapy and recovered

Surgery:

* Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1994-05; Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stan Z. Gertler, MD, FRCPC, Study Chair — Ottawa Regional Cancer Centre
Locations (1):
- Ottawa Regional Cancer Centre at Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Gertler SZ, Yau J, Stewart DJ, et al.: Cisplatin, doxorubicin and tamoxifen (CAT) in the treatment of incurable soft tissue and endocrine malignancies-preliminary results. [Abstract] Proceedings of the American Society of Clinical Oncology 15: A1427, 1996.